CLINICAL TRIAL: NCT06061757
Title: Use of 4D Intracardiac Echocardiography (4D-ICE) in Conjunction With Transesophageal Echocardiography (TEE) for Left Atrial Appendage Closure (LAAC)
Brief Title: Use of 4D-ICE in Conjunction With TEE for Left Atrial Appendage Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KCHRRF_Nuvision ICE_0017
Record Dates: First submitted 2023-09-11; First posted 2023-09-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Echocardiography, Transesophageal; Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1 - TEE Primary imaging guidance (Experimental): TEE is the primary imaging guidance with 4D ICE is the secondary
  Interventions: Device: Imaging guidance with TEE and ICE for Left atrial appendage closure
- Arm 2 - ICE Primary Imaging Guidance (Experimental): 4D ICE is the primary imaging guidance and TEE is the secondary
  Interventions: Device: Imaging guidance with TEE and ICE for Left atrial appendage closure

INTERVENTIONS:
Device: Imaging guidance with TEE and ICE for Left atrial appendage closure — The occluder size for both LAAC devices will be selected based on the maximal diameter of the LAA orifice following the manufacturer guidelines and using the maximal length of the LAA measured on Echocardiogram. Intraprocedural measurements of the LAA width and depth were acquired on both ICE and TEE per protocol. Both ICE and TEE will be used to assess for any procedural complications prior to insertion of the device delivery sheath.

SUMMARY:
This is a prospective, single center, non-randomized study with two parallel arms intended to study if 4D Intracardiac echocardiography (4D-ICE) (Nuvision, Nuvera TM) will provide better visualization of the anatomical landmarks from the larger imaging volume and provide optimal intra procedural guidance similar to Transesophageal echocardiography (TEE) (GE 6VT-D ULTRASOUND TRANSDUCER) for Left atrial appendage closure (LAAC). The study will enroll approximately 52 subjects and will be followed through 12 months.

DETAILED DESCRIPTION:
Standard intraprocedural guidance for transcatheter left atrial appendage closure (LAAC) employs a multi-modality integrated approach combining fluoroscopy for guiding the delivery system, and transesophageal echocardiography (TEE) for intracardiac characterization to guide device selection and monitor procedural complications. Successful implantation of the device is confirmed with contrast-enhanced fluoroscopy and color doppler flow imaging on TEE. TEE is the current gold standard for procedural guidance but requires general anesthesia (GA) to avoid patient motion and discomfort during the procedure. General anesthesia, however, is associated with pulmonary complications and patient discomfort due to endotracheal intubation. Intraprocedural LAAC guidance under local anesthesia or conscious sedation might help mitigate these GA-related disadvantages and has motivated multiple clinical studies, establishing intracardiac echocardiography (ICE) as a safe and feasible alternative to TEE.

The new generation of NuVision ICE catheter offers a larger imaging volume of 90° x 90° with multiplanar reformatted (MPR) echo views for better visualization of anatomical landmarks and procedural guidance and aid in sizing of the device. This has a potential to improve outcomes and reduce procedure times while lowering healthcare costs.

In this study, Role of NuVision Intracardiac Echocardiographic (ICE) catheter with Tranesopheal echocardiography (TEE) in predicting intra-procedural outcomes and success of implantation in patients undergoing left atrial appendage occlusion will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male/Females
* Age:18-80 years
* History of Atrial Fibrillation/Atrial flutter
* Will have endocardial Left Atrial Appendage Closure (LAAC) with an Amplatzer Amulet or WATCHMAN FLX device

Exclusion Criteria:

* Inability or unwillingness of an individual to give written informed consent
* Patient not following with our practice after the procedure
* Complex anatomy for endocardial LAAC
* Thrombus in LAA
* Patients with pericardial effusion in pre-op TEE/CCTA
* Patients currently pregnant (Serum beta HCG completed when labs obtained for the procedure are completed)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Success of Implantation of Left Atrial Appendage Closure (LAAC) device | 1 Day
  Success of Implantation of Amulet or Watchman FLX device

SECONDARY OUTCOMES:
Intraprocedural measurements | 1 Day
  Transeptal access view, LAA thrombus, Stability of the device, Peri-device leaks, Device Repositioning, Clarity of mitral valve or pulmonary vein impingement will be noted as Yes/No from Echocardiogram
Intraprocedural measurements | 1 Day
  LAA size in different sites will be noted from Echocardiograms
Intraprocedural measurements - LAA device size | 1 Day
  LAA device size will be measured based on the LAA size
Location of the leaks | 1 Day
  Location of the leaks will be identified
Intraprocedural measurements | 1 Day
  Procedural duration, Fluoroscopic time

OTHER OUTCOMES:
Post Procedural Outcomes | 45 Days, 6 Months and 12 Months
  Presence of any Peri-device leaks (PDL), Device Related Thrombus (DRTs), Micro migration and device tilt will be noted.
Post Procedural Outcomes - Size of the leaks | 45 Days, 6 Months and 12 Months
  Leaks if any, leaks size will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas, United States

REFERENCES:
- [Background] Sievert H, Lesh MD, Trepels T, Omran H, Bartorelli A, Della Bella P, Nakai T, Reisman M, DiMario C, Block P, Kramer P, Fleschenberg D, Krumsdorf U, Scherer D. Percutaneous left atrial appendage transcatheter occlusion to prevent stroke in high-risk patients with atrial fibrillation: early clinical experience. Circulation. 2002 Apr 23;105(16):1887-9. doi: 10.1161/01.cir.0000015698.54752.6d. PMID 11997272
- [Background] Saw J. Intracardiac Echocardiography for Endovascular Left Atrial Appendage Closure: Is it Ready for Primetime? JACC Cardiovasc Interv. 2017 Nov 13;10(21):2207-2210. doi: 10.1016/j.jcin.2017.07.002. Epub 2017 Aug 30. No abstract available. PMID 28866032
- [Background] Khalili H, Patton M, Taii HA, Bansal P, Brady M, Taylor J, Gurung A, Maini B. 4D Volume Intracardiac Echocardiography for Intraprocedural Guidance of Transcatheter Left Atrial Appendage Closure. J Atr Fibrillation. 2019 Dec 31;12(4):2200. doi: 10.4022/jafib.2200. eCollection 2019 Dec. PMID 32435343
- [Background] Ranard LS, Khalique OK, Donald E, Agarwal V, Hamid N, Hahn RT, Ng V, Brady M, Gurung A, Ali ZA, Leon MB, Sommer R, Vahl TP. Transcatheter Left Atrial Appendage Closure Using Preprocedural Computed Tomography and Intraprocedural 4-Dimensional Intracardiac Echocardiography. Circ Cardiovasc Interv. 2021 Jul;14(7):e010686. doi: 10.1161/CIRCINTERVENTIONS.121.010686. Epub 2021 Jun 23. No abstract available. PMID 34157847
- [Background] http://cardiacvascularnews.com/nuvera-announces-successful-first-in-human-use-of-nuvision-ice-catheter/